CLINICAL TRIAL: NCT03974750
Title: Bimanual Motor Skill Learning Through Robotics in Stroke Survivors and Healthy Individuals
Acronym: bimMsKL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, MD, PhD, Neurologist, Principal Investigator, Clinical Professor, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: bimMsKL
Record Dates: First submitted 2019-05-28; First posted 2019-06-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Evaluation of bimanual motor skill learning Motor skill learning with a rehabilitation robot
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): Training on the rehabilitation robot REAplan(R) to learn complex, coordinated bimanual movements
  Interventions: Device: Bimanual motor skill learning with the REAplan(R) rehabilitation robot
- control intervention (Active Comparator): Training on the rehabilitation robot REAplan(R) with simple movements
  Interventions: Device: Bimanual motor skill learning with the REAplan(R) rehabilitation robot

INTERVENTIONS:
Device: Bimanual motor skill learning with the REAplan(R) rehabilitation robot — REAplan(R) rehabilitation robot : training to perform complex, coordinated, bimanual movements

SUMMARY:
To test the capacity of healthy and chronic stroke patients to learn and retain a complex bimanual motor skill, trained on the neurorehabilitation robot REAplan (R) (bimanual version).

DETAILED DESCRIPTION:
Over 3 consecutive days, healthy individuals and chronic stroke patients (1) will be evaluated and (2) will train on the neurorehabilitation robot REAplan(R).

They will practice several tasks on the robot REAplan (R) (bimanual version), requiring either movements with the affected arm (unimanual tasks) and complex, coordinated movements with both arms (bimanual tasks).

In addition, several "classical" clinical scales and tests will be used to evaluate overall motor-sensory-cognitive functions (clinical tests, questionnaires, ...).

ELIGIBILITY:
STROKE PATIENTS :

Inclusion Criteria:

* having a chronic stroke (>6 months)
* aged 18-90 years
* with demonstrate a stroke lesion on brain imaging.

Exclusion Criteria:

* difficulty in understanding or executing commands
* drug/alcohol abuse
* severe aphasia / cognitive deficits interfering with study
* inability to voluntarily move the affected arm (i.e. complete paralysis of the arm)
* multiple strokes / dementia / psychiatric condition
* botulinum toxin injections (to be evaluated)

HEALTHY INDIVIDUALS :

Inclusion Criteria:

- 18-90 years

Exclusion Criteria:

* neurological conditions interfering with the study
* drug/alcohol abuse
* pyschiatric condition

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
bi-SAT, bimanual Speed/Accurady Trade-off measured by the REAplan robot | change between baseline (Day 1) and after training (Day 3)
  bimanual Speed/Accurady Trade-off: mathematical computation of the relationship bewteen speed and accuracy
bi-CO, bimanual Coordination factor measured by the REAplan robot | change between baseline (Day 1) and after training (Day 3)
  bimanual Coordination factor, mathematical measure of the phase coherence between speeds of both arms
bi-Force, bimanual Coordination factor measured by the REAplan robot | change between baseline (Day 1) and after training (Day 3)
  bimanual forces, forces exerted in the wrong direction by each arm (Newtons)

SECONDARY OUTCOMES:
bi-SAT on bimanual REACHING (REAplan robot) | change between baseline (Day 1) and after training (Day 3)
  bimanual Speed/Accurady Trade-off: mathematical computation of the relationship
bi-Force on bimanual REACHING (REAplan robot) | change between baseline (Day 1) and after training (Day 3)
  bimanual forces, forces exerted in the wrong direction by each arm (Newtons)
bi-CO on bimanual REACHING (REAplan robot) | change between baseline (Day 1) and after training (Day 3)
  bimanual Coordination factor, mathematical measure of the phase coherence between speeds of both arms
bi-smoothness on bimanual REACHING (REAplan robot) | change between baseline (Day 1) and after training (Day 3)
  Smoothness of movement : Spectral Arc Length (SPARC)
bi-error on bimanual REACHING (REAplan robot) | change between baseline (Day 1) and after training (Day 3)
  Error in centimeres or degrees during bimanual reaching
BBT | change between baseline (Day 1) and after training (Day 3)
  Box & Blocks Test (timed transfert of blocks from one space to the other, 3 trials/hand)
whole-hand GF | change between baseline (Day 1) and after training (Day 3)
  whole-hand Grip Force (GF) measured with a dynamometer, 3 trials/hand)
Visual Analog Scale for fatigue (VAS fatigue) | change between baseline (Day 1) and after training (Day 3)
  Visual Analog Scale to evaluate fatigue = a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. Range : 0- 10.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Y Vandermeeren, MD, PhD, Principal Investigator — Université catholique de Louvain, Institute of NeuroScience (IONS) NEUR / CHU
Locations (2):
- Belgium (2):
  - CHU UCL Namur, Mont-Godinne, Neurology Department, Stroke Unit, Yvoir, Namur
  - Department of Neurology, CHU Mont-Godinne, Yvoir, Namur

IPD SHARING:
Plan to Share IPD: Yes
the precise IPD plan has to be worked out in order to find the best public repository
Supporting Information: Study Protocol
Time Frame: Up to 2 years after publication of the scientific articles
Access Criteria: none (public)

REFERENCES:
- [Background] Yeganeh Doost M, Orban de Xivry JJ, Bihin B, Vandermeeren Y. Two Processes in Early Bimanual Motor Skill Learning. Front Hum Neurosci. 2017 Dec 20;11:618. doi: 10.3389/fnhum.2017.00618. eCollection 2017. PMID 29326573
- [Background] Doost MY, Orban de Xivry JJ, Herman B, Vanthournhout L, Riga A, Bihin B, Jamart J, Laloux P, Raymackers JM, Vandermeeren Y. Learning a Bimanual Cooperative Skill in Chronic Stroke Under Noninvasive Brain Stimulation: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2019 Jun;33(6):486-498. doi: 10.1177/1545968319847963. Epub 2019 May 15. PMID 31088342
- [Background] Dehem S, Gilliaux M, Lejeune T, Delaunois E, Mbonda P, Vandermeeren Y, Detrembleur C, Stoquart G. Effectiveness of a single session of dual-transcranial direct current stimulation in combination with upper limb robotic-assisted rehabilitation in chronic stroke patients: a randomized, double-blind, cross-over study. Int J Rehabil Res. 2018 Jun;41(2):138-145. doi: 10.1097/MRR.0000000000000274. PMID 29420360
- [Derived] Gerardin E, Bontemps D, Babuin NT, Herman B, Denis A, Bihin B, Regnier M, Leeuwerck M, Deltombe T, Riga A, Vandermeeren Y. Bimanual motor skill learning with robotics in chronic stroke: comparison between minimally impaired and moderately impaired patients, and healthy individuals. J Neuroeng Rehabil. 2022 Mar 17;19(1):28. doi: 10.1186/s12984-022-01009-3. PMID 35300709
- [Derived] Yeganeh Doost M, Herman B, Denis A, Sapin J, Galinski D, Riga A, Laloux P, Bihin B, Vandermeeren Y. Bimanual motor skill learning and robotic assistance for chronic hemiparetic stroke: a randomized controlled trial. Neural Regen Res. 2021 Aug;16(8):1566-1573. doi: 10.4103/1673-5374.301030. PMID 33433485